CLINICAL TRIAL: NCT06654505
Title: Effectiveness of Village Health Volunteers/Workers Working As Male-Female Pairs on Women's Use of Postnatal Care Services in Sepone District in Lao People's Democratic Republic: a Protocol for a Quasi-experimental Cluster Study
Brief Title: Can Village Health Volunteers/Workers Working As Male-Female Pairs Improve the Use of Postnatal Care Services in the Lao People's Democratic Republic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Ryukyus (Other)
Responsible Party: Principal Investigator, Credo Adelphe Ahissou, Research fellow and Assistant Investigator, University of the Ryukyus
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 24-2329-00-00-00
Record Dates: First submitted 2024-10-15; First posted 2024-10-23 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Pregnant Women; Lactating Mother

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Villages where Village Health Volunteers/Workers work as individuals (No Intervention)
- Villages where Community Health Workers work in pairs (Experimental)
  Interventions: Behavioral: Paired Community Health Workers

INTERVENTIONS:
Behavioral: Paired Community Health Workers — Community Health Workers will promote maternal and child health services as paired female and male
  Arms: Villages where Community Health Workers work in pairs

SUMMARY:
The study aims to assess the effectiveness of male-female VHV/Ws working in pairs on women's uptake of second PNC visits in rural Sepone, Lao PDR.

Methods A quasi-experimental cluster study will be conducted between July 2024 and October 2026 in 37 selected sites from two districts in southern Lao PDR. In 19 selected intervention villages in the Sepone district, female-male VHV/Ws pairs will promote postpartum services, whereas, in 18 similar control villages in the Vilabuly district, VHV/Ws will work as individuals.

ELIGIBILITY:
Inclusion Criteria:

* Women who gave birth within six weeks and twelve months before the study's baseline and end-line surveys.

Exclusion Criteria:

* Women whose births resulted in a loss,
* Women who do consent to participate in the surveys
* Women who face a language barrier with surveyors will not be enrolled.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Only women who delivered a baby within a define period
Enrollment: 302 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of second postnatal care visit | 6 weeks after delivery
  Second postnatal visit within 6 weeks after delivery in a health facility reported in maternal and child health handbook

SECONDARY OUTCOMES:
Lenght of facility-based postpartum stay | cutoff is 12 hours
  Number of hours of stay in health facility after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Sepon and Vilabouly districts, Savannakhet, Laos

IPD SHARING:
Plan to Share IPD: Undecided